CLINICAL TRIAL: NCT00290290
Title: Chlorhexidine-Alcohol Versus Povidone-Iodine for Surgical-Site Antisepsis:A Prospective, Randomized, Multicenter Clinical Trial
Brief Title: Efficacy Study of Antiseptic Preoperative Scrubs in Prevention of Postoperative Infections
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Michael E. DeBakey VA Medical Center (U.S. Federal Agency); Medical College of Wisconsin (Other); US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Rabih Darouiche, Professor of Medicine, Baylor College of Medicine
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: H-14542
Record Dates: First submitted 2006-02-09; First posted 2006-02-13 (Estimated); Results first posted 2014-08-11 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2014-09

CONDITIONS: Postoperative Wound Infection
Keywords: Prevention; Antiseptic Preoperative Scrub; Postoperative Wound Infection
MeSH Terms: conditions — Surgical Wound Infection | interventions — Chlorhexidine; Ethanol; Povidone-Iodine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- povidone-iodine (Active Comparator): preoperative skin preparation with povidone-iodine
  Interventions: Drug: Povidone-Iodine
- chlorhexidine-alcohol (Experimental): preoperative skin preparation with scrub and paint technique
  Interventions: Drug: chlorhexidine-alcohol

INTERVENTIONS:
Drug: chlorhexidine-alcohol — Preoperative skin preparation with scrub and paint technique
  Other Names: Chloraprep
  Arms: chlorhexidine-alcohol
Drug: Povidone-Iodine — preoperative skin preparation with scrub and paint technique
  Other Names: Betadine
  Arms: povidone-iodine

SUMMARY:
Most cases of infection of clean-contaminated wounds (wounds without gross spillage of organisms from the gastrointestinal tract) are thought to originate from the skin. Therefore, it is conceivable that application of an optimal antiseptic agent can reduce the rate of surgical wound infections. This trial is to compare the impact of disinfecting the skin with Chloraprep (2%chlorhexidine and 70% isopropyl alcohol) vs. Betadine on the rates of infection of clean-contaminated surgical wounds. The study will also assess the occurrence of adverse effects on the skin from either antiseptic agent and the cost-savings associated with the use of Chloraprep vs Betadine.

DETAILED DESCRIPTION:
This is a prospective, randomized, multicenter clinical trial. All adult patients, who are scheduled for a clean-contaminated surgical procedure of the alimentary, respiratory, reproductive or urinary tract will be asked to participate.

ELIGIBILITY:
Inclusion Criteria: Adult patients who are scheduled for a clean-contaminated surgical procedure of the alimentary or respiratory tract will be eligible for participation. A clean-contaminated wound is one that is entered under controlled conditions without unusual contamination.

-

Exclusion Criteria: Patients will be excluded form the study if: (1) they are unable or unwilling to give informed consent; (2) the patient is less than 18 years of age; (3) there is evidence of pre-existing infection at or adjacent to the operative site; (4) a break in sterile technique occurs; (5) the patient has a history of allergy to chlorhexidine, alcohol or iodophors.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 849 (Actual)
Dates: Start 2003-09; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rabih O Darouiche, M.D., Study Chair — Baylor College of Medicine
Locations (6):
- United States (6):
  - Veterans Affairs Boston Healthcare System, West Roxbury, Massachusetts
  - Durham VA Medical Center, Durham, North Carolina
  - Ben Taub General Hospital, Houston, Texas
  - Michael E Debakey Medical Center, Houston, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Milwaukee VA Medical Center, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Darouiche RO, Wall MJ Jr, Itani KM, Otterson MF, Webb AL, Carrick MM, Miller HJ, Awad SS, Crosby CT, Mosier MC, Alsharif A, Berger DH. Chlorhexidine-Alcohol versus Povidone-Iodine for Surgical-Site Antisepsis. N Engl J Med. 2010 Jan 7;362(1):18-26. doi: 10.1056/NEJMoa0810988. PMID 20054046

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients 18 years or older undergoing clean-contaminated surgery preformed without substantial spillage or unusual contamination were eligible for enrollment. Patients were excluded if they were allergic to chlorhexidine, alcohol, or iodophors, or had infection at or adjacent to operative site, & if there was a perceived inability for a 30 days F/U
Pre-assignment Details: There were no significant events prior to group assignment. Enrolled patients were immediately and randomly assigned in a 1:1 ratio to a study arm. To help match the two groups and address potential inter-hospital differences, randomization was stratified by hospital with the use of computer-generated randomization numbers without blocking
Groups:
- Povidone-Iodine: Skin at surgical site preoperatively scrubbed then painted with an aqueous solution of 10% povidone-iodine
- Chlorhexidine-Alcohol: Skin at surgical site preoperatively scrubbed with an applicator that contained 2% chlorhexidine gluconate and 70% alcohol
Period: Overall Study
Arm/Group | Povidone-Iodine | Chlorhexidine-Alcohol
Started | 440 | 409
Completed | 422 | 391
Not Completed | 18 | 18
Not completed — Death | 3 | 4
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Underwent clean surgical procedure | 13 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Povidone-iodine | Chlorhexidine-alcohol | Total
Number analyzed (Participants) | 440 | 409 | 849
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.9 (14.2) | 53.3 (14.6) | 53.1 (14.4)
Age, Customized [Number; unit: participants]
  <18 years | 0 | 0 | 0
  >18 years | 440 | 409 | 849
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 194 | 168 | 362
  Male | 246 | 241 | 487
Region of Enrollment [Number; unit: participants]
  United States | 440 | 409 | 849

OUTCOME MEASURES:

1. Primary Outcome: The Primary Objective of This Trial is to Compare the Impact of Disinfecting the Skin With Chloraprep vs. Betadine on the Rates of Infection of Clean-contaminated Surgical Wounds.
Description: The primary end point of the study was the occurrence of any surgical-site infection. Diagnosis of surgical-site infection was diagnosed by a blinded reviewer following criteria developed by the Center for Disease Control. The significance of difference between the two study groups in terms of patient characteristics was determined with the use of the Wilcoxon rank-sum test for continuous variables and Fisher's exact test for categorical variables. For efficacy outcomes, we compared the proportions of patients in the two study groups who could be evaluated and who any type of surgical-site infection using Fisher's exact test and calculating the relative risk of infection and 95% confidence intervals. To determine whether the results were consistent across the 6 participating hospitals, a prespecified Breslow-Day test for homogeneity was performed.
Time Frame: during surgery and within the 30 days post surgery
Measure: Number; unit: Percentage of Post Operative Infections
Arm/Group | Povidone-Iodine | Chlorhexidine-Alcohol
Number analyzed (Participants) | 440 | 409
Percentage of Post Operative Infections | 16.1 [0.41 to 0.85] | 9.5 [0.41 to 0.85]
Statistical Analysis 1: Comparison: Povidone-Iodine vs Chlorhexidine-Alcohol; The average baseline rate of surgical-site infection at the six participating hospitals was 14% after clean-contaminated surgery with povidone-iodine skin preparation, and we estimated that substituting chlorhexidine-alcohol for povidone-iodine would reduce this rate to 7%. Therefore, we planned to enroll approximately 430 patients in each study group who could be evaluated in order for the study to have 90% power to detect a significant difference in the rates of surgical-site infection; Test type: Superiority or Other; p = 0.004, Log Rank; Relative Risk = 0.59, 95% CI 2-sided [0.41 to 0.85]

ADVERSE EVENTS:
Arm/Group | Povidone-Iodine | Chlorhexidine-Alcohol
Serious Adverse Events (participants affected / at risk) | 3/440 | 4/409
Other Adverse Events (participants affected / at risk) | 3/440 | 3/409
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Povidone-Iodine (N=440) | Chlorhexidine-Alcohol (N=409)
Death (Surgical and medical procedures) | 3 (3) | 4 (4) — Death was NOT judged to be related to the study drugs in either group.
OTHER ADVERSE EVENTS (reported when occurring in more than 0.7% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Povidone-Iodine (N=440) | Chlorhexidine-Alcohol (N=409)
Pruritis/Erythema (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No